CLINICAL TRIAL: NCT01290575
Title: Placebo-Controlled, Ascending Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-820132 in Subjects With Type 2 Diabetes Treated With Metformin Monotherapy.
Brief Title: Multiple Ascending Dose Study of BMS-820132 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB122-004
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Arm 1 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 2 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 3 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 4 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 5 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 6 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 7 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 8 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132
- Arm 9 BMS-820132 or placebo (Active Comparator)
  Interventions: Drug: Placebo; Drug: BMS-820132

INTERVENTIONS:
Drug: Placebo — capsule, Oral, 0.0mg, twice daily, 14 day
  Arms: Arm 1 BMS-820132 or placebo; Arm 2 BMS-820132 or placebo; Arm 3 BMS-820132 or placebo; Arm 4 BMS-820132 or placebo; Arm 5 BMS-820132 or placebo; Arm 9 BMS-820132 or placebo
Drug: Placebo — Capsule, Oral, 0.0mg, once daily, 14 day
  Arms: Arm 6 BMS-820132 or placebo; Arm 7 BMS-820132 or placebo; Arm 8 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, 15mg, twice daily, 14 day
  Arms: Arm 1 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, 60mg, twice daily, 14 day
  Arms: Arm 2 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, oral, 150mg, twice daily, 14 day
  Arms: Arm 3 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, 300mg, twice daily, 14 day
  Arms: Arm 4 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, 450mg, twice daily, 14 day
  Arms: Arm 5 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, To be determined (TBD), once daily, 14 day
  Arms: Arm 6 BMS-820132 or placebo; Arm 7 BMS-820132 or placebo; Arm 8 BMS-820132 or placebo
Drug: BMS-820132 — Capsule, Oral, 5 mg, twice daily, 14 day
  Arms: Arm 9 BMS-820132 or placebo

SUMMARY:
BMS-820132 is an investigational new drug being developed by BMS for treating Type 2 diabetes. The purpose of this study is to test the safety/tolerability (potential side effects) of multiple doses of the investigational new drug, as well as the amount of study drug in the blood and its effects on blood sugar,in subjects with type 2 diabetes.

DETAILED DESCRIPTION:
Study Classification: Safety, Pharmacokinetics/dynamics

ELIGIBILITY:
Inclusion Criteria:

* Males and females of childbearing potential (willing to use an acceptable method of contraception), or females of non-childbearing potential (i.e., post-menopausal or surgically sterile).
* Diagnosis of type 2 diabetes treated with metformin monotherapy (at least 1500 mg/day for at least 6 months) on a stable regimen for at least 2 months.
* Body Mass Index (BMI) of 18.5 to 40 kg/m2.
* Fasting glucose in the range of 125-275 mg/dL.
* Hemoglobin A1c (HbA1c) in the range of 7.0% -11.0%.
* Fasting C-peptide > 1 ng/mL.

Exclusion Criteria:

* Clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations, and any significant acute or chronic medical illness other than stable and well controlled hypertension, microalbuminuria, dyslipidemia, depression, or hypothyroidism.
* History of diabetic ketoacidosis, hyperosmolar nonketotic syndrome, lactic acidosis, hypoglycemia (i.e., ≥ 1 self-reported episodes of hypoglycemia within the last 3 months or ≥ 2 self-reported episodes of hypoglycemia within the last 6 months), or hypoglycemia unawareness.
* Any major surgery within 4 weeks of study drug administration.
* Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Smoking more than 10 cigarettes per day.
* Recent drug or alcohol abuse.
* Women who are pregnant or breastfeeding.
* Positive urine screen for drugs of abuse.
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus (HIV)-1, -2 antibody.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Adverse events, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments. | Throughout the study drug administration period (14 days)
Adverse events, physical examinations, clinical laboratory determinations, electrocardiograms (ECG), and vital sign assessments. | within 7 days after the final dose

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-820132 | Day 1 and Day 14
Time of maximum observed plasma concentration (Tmax) of BMS-820132 | Day 1 and Day 14
Trough observed plasma concentration (Cmin) of BMS-820132 | Day 1 through Day 14 (selected days)
Area under the plasma concentration-time curve over one dosing interval [AUC(TAU)] of BMS-820132 | Day 1 and Day 14
Accumulation index (AI) of BMS-820132 | Day 14
Half life (T-Half) of BMS-820132 | Day 14
AUC(0-24 h) and postprandial AUC(0-4h) for biomarkers of glucose homeostasis | Day -1, Day 1, Day 7 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Dedicated Phase I, Inc., Phoenix, Arizona
  - Osborne Research Center, Little Rock, Arkansas
  - Clinical Pharmacology Of Miami Inc., Miami, Florida
  - Mra Clinical Research, Miami, Florida
  - Cetero Research, San Antonio, Texas

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx